CLINICAL TRIAL: NCT07147595
Title: Chronic Effect of Isometric Exercise on Blood Pressure in Patients With Controlled Hypertension: a Randomized Clinical Trail
Brief Title: Chronic Effect of Isometric Exercise on Blood Pressure in Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Patricia Caetano, PhD student, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UP5965-21
Record Dates: First submitted 2025-08-14; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hypertension (HTN); Hypertension Arterial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Isometric handgrip exercise (Experimental): Small Mass Muscle - isometric handgrip exercise
  Interventions: Procedure: Isometric handgrip exercise
- Isometric knee extension exerice (Experimental): Large Mass Muscule - isometric knee extension exercise
  Interventions: Procedure: Isometric knee extension exercise

INTERVENTIONS:
Procedure: Isometric handgrip exercise — Participants will train 3 times per week for 4 weeks. Each session will consist of four sets of 2-minute contractions sustained at 30% of maximum voluntary contraction (MVC), performed with a handgrip device for each arm, with 1-minute rest intervals between sets and between arms.
  Arms: Isometric handgrip exercise
Procedure: Isometric knee extension exercise — Participants will train 3 times per week for 4 weeks. Each session will consist of four sets of 2-minute contractions sustained at 30% of maximum voluntary contraction (MVC), performed with adjustable ankle weights for each leg, with 1-minute rest intervals between sets and between legs.
  Arms: Isometric knee extension exerice

SUMMARY:
International recommendations support dynamic or isometric strength training as an adjunct to aerobic exercise. Given the lack of consensus, this study aims to evaluate the chronic effects of isometric exercise, performed through handgrip or isometric knee extension, as a hypotensive strategy in adults with hypertension.

DETAILED DESCRIPTION:
This study is designed as a randomized, controlled, evaluator-blinded clinical trial, conducted entirely at the Laboratory of Clinical Investigation (LCI) of the Cardiology Institute of Rio Grande do Sul / University Foundation of Cardiology (ICFUC). The project follows all recommendations of the CONSORT Statement.

Male and female participants aged 40 to 70 years, with blood pressure ≥ 120/80 mmHg, will be enrolled. After signing informed consent, participants will complete a questionnaire to assess their habitual physical activity level and will undergo isometric handgrip or isometric knee extension training for 4 weeks. Blood pressure will be assessed at baseline and after the intervention using ambulatory blood pressure monitoring (ABPM).

ELIGIBILITY:
Inclusion Criteria:

Patients with controlled hypertension under medication. Sedentary or physically inactive individuals.

Exclusion Criteria:

Pregnant women. Unstable angina. Heart failure classified as NYHA class II, III, or IV. Recent cardiovascular event within the last 3 months. Chronic renal insufficiency. Diabetes mellitus. History of malignant disease with a life expectancy of less than 2 years. Orthopedic, physical, or mental limitations that prevent the performance of physical exercise.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Bood pressure | Assessments (systolic/diastolic pressure) will be performed at baseline and after 4 weeks of training (post-intervention).
  Bood pressure (systolic and diastolic) measured by Ambulatory Blood Pressure Monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Lehnen, PhD, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No